CLINICAL TRIAL: NCT02686697
Title: A Double-blind, Placebo-controlled Study on the Effects of Combined L-Carnosine and Cognitive Training on Cognition in Schizophrenia
Brief Title: Carnosine and Cognitive Training in Schizophrenia
Acronym: CACTIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abraham Reichenberg (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Abraham Reichenberg, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 14-1119
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
Keywords: L-Carnosine; Schizophrenia; Psychosis; Cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Carnosine; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Carnosine (Experimental): oral doses of 2000mg for 4 weeks total - 2 weeks medication phase only, and then 2 weeks combined treatment with cognitive training.
  Interventions: Drug: L-Carnosine; Behavioral: Cognitive Training
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo; Behavioral: Cognitive Training

INTERVENTIONS:
Drug: L-Carnosine
  Other Names: Carnosine
  Arms: L-Carnosine
Drug: Placebo
  Arms: Placebo
Behavioral: Cognitive Training — Cognitive Training for 2 weeks

SUMMARY:
This is a double-blind placebo-controlled trial to evaluate the effects of the combination of a cognition enhancing drug, i.e carnosine, with cognitive training in patients with schizophrenia. All participants will receive the same cognitive training sessions and will be randomised to either carnosine or placebo for the duration of the combined treatment period (2 weeks). Before combined training and carnosine/placebo, there is a two-week carnosine/placebo only phase to examine the effects of carnosine alone on functioning without training.

DETAILED DESCRIPTION:
Compromised cognitive functioning is a core feature of schizophrenia, yet it remains a major unmet need in the treatment of schizophrenia. Current available therapeutic approaches to enhance cognition in schizophrenia - either pharmacological or non-pharmacological (for a review) have yielded, at best, only modest results with questionable retention of the cognitive benefits and generalization of the effects into functional benefit. The investigators propose a novel approach to enhance cognition in schizophrenia: combining a food supplement with cognitive training, rather than using each intervention alone.

Aim is to test the primary hypothesis that the combination of L-carnosine with cognitive training will significantly increase the performance of patients with schizophrenia on memory and learning training tasks compared to pairing cognitive training with placebo. The investigators will also test the secondary hypotheses that in the group receiving L-carnosine increased performance is due to a greater learning rate. Carnosine has antioxidant and antiglycating action and is found in food and the human body. The investigator's choice is guided by several considerations but, primarily the evidence that L-carnosine has neuroprotective effects through its antioxidant features. Briefly, the investigators propose that alterations in metabolism in several neurotransmitter systems (particularly glutamate) can both contribute to, and be modified by, oxidative stress, and therefore antioxidant administration could positively affect neurotransmitter role in synaptic plasticity, learning and memory.

Carnosine has shown some improvements in cognitive outcomes in autism (Chez et al, 2002) and schizophrenia (Chengappa et al; unpublished). Chez used oral doses of 800mg/d for 8 weeks; while the latter study used oral doses of 2000mg for 4 weeks showing positive effects. Hence this is the dose and delivery route that will be used. The investigators have opted for 4 weeks course following broadly from these two studies. Carnosine is widely available from health and food supplement shops in the UK and US retail market in highly pure form; is a naturally occurring in food and the human body; and is well-tolerated and has a benign side-effect profile, as shown from previous trials, and is therefore not associated with any potential risks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60, males and females.
* DSM-IV diagnosis of schizophrenia or schizoaffective disorder documented in a medical record, confirmation by treating physician and/or treatment team, or confirmation of diagnosis by our study psychiatrist or clinical psychologist
* Duration of illness equal to or greater than one year.
* Patients should be clinically stable in a non-acute phase for at least 8 weeks prior to the screening visit
* Treatment with stable doses of antipsychotic medications for at least 4 weeks prior to the screening visit.
* Negative result in the urine pregnancy test performed during the screening visit in women of child bearing potential (not surgically sterile or 2 years postmenopausal).Women of child-bearing potential, who are sexually active, will be considered as potential participants if they are using acceptable methods of contraception, which include barrier method with spermicide, intrauterine device (IUD), steroidal contraceptive (oral, transdermal, implanted, and injected).
* Subjects must read and write in English at a level sufficient to understand and complete study- related procedures.
* Informed consent signed by participant

Exclusion Criteria:

* DSM -IV diagnosis of alcohol or substance abuse (other than nicotine) within the last month or a DSM-IV]diagnosis of alcohol or substance dependence (other than nicotine) in the last 6 months preceding the screening visit.
* Current treatment (within 4 weeks) with psychotropic agents known to effect cognition: amphetamines, barbiturates, MAOIs, methylphenidate, benzodiazepines.
* Pregnant or breast-feeding women.
* Clinically significant abnormalities on physical examination.
* History of a serious neurological disorder or a systemic illness with known neurological complications.
* History of significant other major or unstable metabolic, hepatic, renal, hematological, pulmonary or cardiovascular disorders.
* Known allergy to L-carnosine
* Unwillingness or inability to follow or comply with the procedures outlined in the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Cognitive Training Score | 8 weeks
  Cognitive Training Score will test whether the combination of L-carnosine with cognitive training will significantly increase the performance of patients with schizophrenia on memory and learning training tasks compared to pairing cognitive training with placebo.

SECONDARY OUTCOMES:
The Learning Rate | 8 weeks
  The Learning Rate will test whether the group receiving L-carnosine increased performance is due to a greater learning rate.
Change in Performance Advantage | 8 weeks and 10 weeks
  Performance Advantage will test whether performance advantage is retained after cessation of L-carnosine and training, contrary to a state-dependent effect. Compares performance between week 10 and week 8. An advantage (if exists) is a difference between the treatment arm and the placebo arm of the trial on the primary outcome measure. For an advantage the treatment arm should perform better than the placebo arm. If there is no difference between the groups or that the placebo group performs better than the treatment group than the treatment offers no advantage.
Matrix Consensus Cognitive Battery (MCCB) | 8 weeks
  MCCB composite score will test whether the enhanced learning on specific tasks will generalize into enhanced performance

CONTACTS AND LOCATIONS:
Overall Officials: Avi Reichenberg, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States